CLINICAL TRIAL: NCT06864949
Title: Efficacy of Transverse Maxillary Expansion With AMCOP Preformed Appliances: Prospective Clinical Study
Brief Title: Efficacy of Transverse Maxillary Expansion With AMCOP Preformed Appliances
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-AMCOP
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Transverse Maxillary Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with AMCOP First Class appliance (Experimental)
  Interventions: Device: AMCOP appliance

INTERVENTIONS:
Device: AMCOP appliance — The device measure will be determined with OrthoCad program on digital models, taking the distance between the vestibular cusps of the upper first molars, at the level of the most prominent point. AMCOPs are preformed devices and there are five different measures based on transverse diameter: 1 (45mm), 2 (50mm), 3 (55mm), 4 (60mm), 5 (65mm).
  Requiring expansion, we will choose an higher AMCOP measure than the transverse distance measured on the digital models at T0.
  The clinical indications for use of the AMCOP device will be as follow:
  * in the first week, wear the appliance during the night and for 30 minutes during the day
  * from the second week onward, wear the appliance for one hour during the day and throughout the night During this time, every month we will visit patients and we will expand the device by soaking it in hot water at about 70 °C for 30 s and then in cold water to stabilize it in its new shape.

SUMMARY:
The present study aimed to investigate the cross-sectional effect of Class I AMCOP devices in patients of all possible skeletal types from both vertical skeletal pattern (normodivergent, hyperdivergent, hypodivergent) and sagittal skeletal pattern (skeletal Class I, skeletal Class II, skeletal Class III).

The criterion for choosing patients was determined by the protocol of using these devices, which is to always perform an AMCOP First Class phase with the aim of improving transverse coordination of the arches, Spee's Curve and Wilson's Curve.

DETAILED DESCRIPTION:
This prospective clinical study will investigate the cross-sectional effect of Class I AMCOP (Cranium Occluded Postural Multifunctional Harmonizers, Micerium spa) devices in patients of all possible skeletal types from both vertical skeletal pattern (normodivergent, hyperdivergent, hypodivergent) and sagittal skeletal pattern (skeletal Class I, skeletal Class II, skeletal Class III).

Patients willing to start AMCOP therapy and recruited for the study will be asked to sign the informed consent. Parents will sign the consent for underage patients.

We will recruit patients by following specific inclusion and exclusion criteria during an orthodontic examination.

Diagnostic records will be recorded before treatment (T0) and after 10-12 months of treatment (T1) and included:

* Intraoral and extraoral photographs
* Impressions of the dental arches with digital scanner
* Orthopantomography
* Lateral teleradiography

Changes will be evaluated at T0 and T1 as follows:

* cross-sectional effects will be analyzed on digital models of the upper and lower arch, taking the following linear measurements with OrthoCad program:

  1. upper and lower intermolar distance (taking as reference the top of the mesiovestibular cusp of the upper first molars)
  2. upper and lower intercanine distance (taking as reference the top of the cusp)
* skeletal changes in latero-lateral teleradiography will be analyzed by using "Giannì cephalometric analysis" The expected duration of the first phase of therapy is averaged 10-12 months. During this time, every month patients will be visited and the devices will be activated.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting maxillary transverse deficits (that includes: posterior crossbite monolateral or bilateral; end-to-end occlusal relationships; excessive linguoinclination of lower posterior teeth due to the contraction of maxillary arch; limited permutation space of permanent elements)
* patients with all sagittal and vertical skeletal patterns

Exclusion Criteria:

* syndromic patterns, cleft lip or cleft palate, severe malformations of the maxillae, severe skeletal asymmetry
* physical or psychological limitations
* presence of metallic restorations
* previous orthodontic treatments

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in upper intermolar distance on digital casts | Before treatment (T0) and after 10-12 months of treatment (T1)
  The upper intermolar distance take as reference the top of the mesiovestibular cusp of the upper first molars.

SECONDARY OUTCOMES:
Change in upper intercanine distance on digital casts | Before treatment (T0) and after 10-12 months of treatment (T1)
  The upper intercanine distance take as reference the top of upper canine cusp.
Change in lower intercanine distance on digital casts | Before treatment (T0) and after 10-12 months of treatment (T1)
  The lower intercanine distance take as reference the top of lower canine cusp.
Change in ANB angle | Before treatment (T0) and after 10-12 months of treatment (T1)
  ANB angle will be calculated using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Wits Index | Before treatment (T0) and after 10-12 months of treatment (T1)
  Wits Index will be calculated using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Skeletal Class | Before treatment (T0) and after 10-12 months of treatment (T1)
  Skeletal Class will be assessed combining the ANB angle and Wits Index values using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Cranio-Mandibular Angle | Before treatment (T0) and after 10-12 months of treatment (T1)
  Cranio-Mandibular Angle will be evaluated between SN and GoGn planes following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Intermaxillary Angle | Before treatment (T0) and after 10-12 months of treatment (T1)
  Intermaxillary Angle will be evaluated between bispinal and mandibular planes following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Skeletal Vertical Pattern: | Before treatment (T0) and after 10-12 months of treatment (T1)
  Skeletal vertical pattern will be assessed using Cranio-Mandibular and Intermaxillary Angles following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Articular Angle | Before treatment (T0) and after 10-12 months of treatment (T1)
  Articular Angle will be evaluated between SArGo points following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Upper and Lower Goniac Angles | Before treatment (T0) and after 10-12 months of treatment (T1)
  Upper and Lower goniac angles will be evaluated between respectively Ar-Go-N and N-Go-Gn points following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Mandibular growth pattern | Before treatment (T0) and after 10-12 months of treatment (T1)
  Mandibular growth pattern will be assessed using Articular Angle and Upper and Lower Goniac Angles, following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Upper incisors Inclination | Before treatment (T0) and after 10-12 months of treatment (T1)
  Upper incisors Inclination will be evaluated between upper incisors Axis and bispinal plane, following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Lower incisors Inclination | Before treatment (T0) and after 10-12 months of treatment (T1)
  Upper incisors Inclination will be evaluated between lower incisors Axis and mandibular plane, following Giannì analysis and using the pre-treatment and the post-treatment lateral cephalometric radiographs.
Change in Dento-alveolar discrepancy | Before treatment (T0) and after 10-12 months of treatment (T1)
  Dento-alveolar discrepancy will be calculated using the pre-treatment and the post-treatment study models using "Tanaka and Jhonston" space Analysis
Change in lower intermolar distance | Before treatment (T0) and after 10-12 months of treatment (T1)
  The lower intermolar distance take as reference the top of the mesiovestibular cusp of the lower first molars.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.